CLINICAL TRIAL: NCT01382576
Title: Women With Polycystic Ovary Syndrome Have Increased Plasma Chitotriosidase Activity: A Pathophysiological Link Between Inflammation and Impaired Insulin Sensitivity?
Brief Title: Women With Polycystic Ovary Syndrome Have Increased Plasma Chitotriosidase Activity
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Aydogan Aydogdu, MD, Gulhane School of Medicine
Other Study IDs: 1491-81-11/1539-1563; Chitotriosidase activity (Other Grant/Funding Number: 1202-0811)
Record Dates: First submitted 2011-06-10; First posted 2011-06-27 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2010-12

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; chitotriosidase activity
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — No biospecimens were to be retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PCOS patients
- PCOS patients and healthy controls: There are two groups in this study. One group is PCOS patients and other group is healthy controls.

SUMMARY:
In the present study, serum chitotriosidase activity and its relationship with insulin resistance were determined in patients with Polycystic Ovary Syndrome (PCOS).

DETAILED DESCRIPTION:
ChT activity is increased in patients with PCOS in concordance with insulin resistance. These findings may reflect the pronounced risk for metabolic syndrome and atherosclerotic diseases in this particular patient group.

ELIGIBILITY:
Inclusion Criteria:

* Absence of significant abnormalities on physical examination except hirsutism
* no lipid lowering, hypoglycemic, antihypertensive or hormone replacement therapy
* normal thyroid function and prolactin level
* absence of history or evidence of metabolic, cardiovascular, respiratory or hepatic disease

Exclusion Criteria:

* Pregnant
* ovarian tumors
* congenital adrenal hyperplasia or BMI greater than 30 kg/m2

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 34 women with PCOS and 44 healty women as control group.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aydogan Aydogdu, MD, Principal Investigator — No organizational affiliation
Locations (1):
- Gulhane School of Medicine Etlik, Ankara, Turkey (Türkiye)